CLINICAL TRIAL: NCT06229717
Title: Vestibular ASsessment In Children - Balance Function in Normal Children and Specific Risk Groups (VASIC)
Brief Title: Vestibular and Postural Function in an Unselected Group of Children With Sensorineural Hearing Loss
Acronym: VASIC
Status: Recruiting | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Principal Investigator, Signe Fiil Bønløkke, Principal Investigator, Gødstrup Hospital
Other Study IDs: SFB-3-2023
Record Dates: First submitted 2024-01-08; First posted 2024-01-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Children, Only; Vestibular Disorder; Vestibular Function; Sensorineural Hearing Loss
Keywords: Vestibular dysfunction; Balance problem; Children; Hearing Loss; Dizziness; Vestibular assessment; video Head Impulse Test; Vestibular Evoked Myogenic Potential; Computerized Dynamic Posturography; Quality of life
MeSH Terms: conditions — Vestibular Diseases; Hearing Loss, Sensorineural; Hearing Loss; Dizziness | interventions — Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with sensorineural hearing loss: Children in the age of 3-10 years with either unilateral or bilateral sensorineural hearing loss is recruited at The Audiologic Clinic at Viborg Regional Hospital, Denmark
  Interventions: Diagnostic Test: video Head Impulse Test; Diagnostic Test: Cervical Vestibular Evoked Myogenic Potential; Diagnostic Test: Ocular Vestibular Evoked Myogenic Potential; Diagnostic Test: Computerized Dynamic Posturography; Other: Dizziness Handicap Inventory for patient caregivers

INTERVENTIONS:
Diagnostic Test: video Head Impulse Test — For v-HIT, the Synapsys v-HIT Ulmer device is used.
  Other Names: vHIT
Diagnostic Test: Cervical Vestibular Evoked Myogenic Potential — For cVEMP, the Eclipse (Interacoustic, Middelfart, Denmark) is used. To bypass the frequent middle ear problems bone conduction stimuli (B-81, Interacoustic, Middelfart, Denmark) are administrated. The bone conductor is placed on the mastoid process and two trials at 70 dB nHL are conducted to check waveform reproducibility. 500 Hz short tone bursts (2-2-2 ms) are applied at 5 per second stimulus repetition rate.
  Other Names: cVEMP
Diagnostic Test: Ocular Vestibular Evoked Myogenic Potential — For oVEMP, the Eclipse (Interacoustic, Middelfart, Denmark) is used. To bypass the frequent middle ear problems bone conduction stimuli (B-81, Interacoustic, Middelfart, Denmark) are administrated. The bone conductor is placed on the mastoid process and two trials at 70 dB nHL are conducted to check waveform reproducibility. 500 Hz short tone bursts (2-2-2 ms) are applied at 5 per second stimulus repetition rate.
  Other Names: oVEMP
Diagnostic Test: Computerized Dynamic Posturography — To evaluate functional balance of the children and the relative contributions of the vision, proprioception, and vestibular system a CDP from Virtualis (Virtualis, Montpellier, France) is used.
  Other Names: CDP
Other: Dizziness Handicap Inventory for patient caregivers — DHI is a caregiver-reported 21- item questionnaire. It is designed to evaluate the perceived quality of life and handicap resulting from dizziness and unsteadiness for the pediatric population. For each question there are three possible answers: yes, sometimes or no. Each answer provides respectively 4, 2 and 0 points. The total DHI scores range from 0 to 84 with higher score being consistent with more limitation and more severe handicap. Scores under 16 are characterized as no limitation or handicap. A score from 16-26 present a mild perceived handicap and mild limitations. A DHI-score between 26-43 is classified as a moderate problem, and a score above 43 describes a severe perceived handicap and severe limitations.
  Other Names: DHI-PC

SUMMARY:
The goal of this prospective cohort study is to investigate the vestibular function in children with unilateral or bilateral sensorineural hearing loss. The main hypothesis of the study is that abnormal vestibular test results will be found in 20-30 % of the children with sensorineural hearing loss. The participants will be children in the age of 3-10 years with sensorineural hearing loss. The test protocol consists of questionnaires and vestibular and postural assessments.

DETAILED DESCRIPTION:
Balance problems in children are an overlooked issue in the Danish healthcare system. Dysfunction of the vestibular system, i.e. vestibular dysfunction (VD), can have significant consequences for children's development and quality of life.

In particular, children with sensorineural hearing loss are at risk of developing VD. Hence, VD has been reported in 14 % to 91 % of children with sensorineural hearing loss. The close anatomical and embryological relationship between the hearing system and the vestibular system may of course explain this correlation.

The investigators aim for a child friendly and reliable vestibular test protocol in the study. According to the investigators studies as well as international reports, the investigators have chosen a vestibular test protocol with Video Head Impulse Test (v-HIT), cervical and ocular Vestibular Evoked Myogenic Potential (c and oVEMP) as the tests are feasible, valid, and child friendly. To evaluate overall balance ability, the children are tested on a Computerized Dynamic Posturography.

The aim of the study is to investigate the vestibular function in children with unilateral or bilateral sensorineural hearing loss.

Hypothesis: The investigators expect that abnormal vestibular test results will be found in 20-30 % of the children with sensorineural hearing loss.

Methods: The study is a prospective cohort study. Participants are a prospective, unselected group of children in the age of 3-10 years with either unilateral or bilateral sensorineural hearing loss. The participants are recruited at The Audiologic Clinic at Viborg Regional Hospital, Denmark.

All participants will go through a test protocol consisting of questionnaires and vestibular and postural assessments.

The primary endpoints are results of v-HIT, c and oVEMP, and posturography, which are compared to normative values. The secondary endpoints are prevalence of vestibular dysfunction and mean total Dizziness Handicap Inventory for patient caregivers (DHI-PC) score. A number of variables are collected such as demographics, developmental milestones, family history with focus on hearing and balance.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age of 3-10 years
* Uni- or bilateral sensorineural hearing loss > 20 dB bone conduction pure tone average measured at frequencies 0.5, 1, 2, 4 kHz
* Written informed consent from the parents.

Exclusion Criteria:

* Previous inner ear surgery
* Visual impairment to such a degree that the child is not able to maintain fixation on a dot one meter away.
* Congenital nystagmus
* Compromised eye muscle mobility
* VEMP-electrode allergy
* History of symptomatic head or neck trauma
* Prescription of medicine which alters vestibular outputs (for instance sedative antihistamines)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A prospective, unselected group of children in the age of 3-10 years with either unilateral or bilateral sensorineural hearing loss is recruited at The Audiologic Clinic at Viborg Regional Hospital, Denmark. We intend to include all consecutive children fitting the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
video Head Impulse Test (vHIT) | Measured at baseline.
  Outcome measures: mean VOR gain
video Head Impulse Test (vHIT) | Measured at baseline.
  Outcome measures: VOR gain asymmetry in percent (%)
video Head Impulse Test (vHIT) | Measured at baseline.
  Outcome measures: description of saccades (overt and covert saccades)
Cervical Vestibular Evoked Myogenic Potential (cVEMP): | Measured at baseline.
  Outcome measures: latency P1 and latency N1 in milliseconds (ms)
Cervical Vestibular Evoked Myogenic Potential (cVEMP): | Measured at baseline.
  Outcome measures: rectified interpeak amplitude P1-N1
Cervical Vestibular Evoked Myogenic Potential (cVEMP): | Measured at baseline.
  Outcome measures: averaged EMG in μV
Cervical Vestibular Evoked Myogenic Potential (cVEMP): | Measured at baseline.
  Outcome measures: left-right asymmetry ratio in percent (%)
Ocular Vestibular Evoked Myogenic Potential (oVEMP): | Measured at baseline.
  Outcome measures: latency N1 and latency P1 in milliseconds
Ocular Vestibular Evoked Myogenic Potential (oVEMP): | Measured at baseline.
  Outcome measures: interpeak amplitude N1-P1 in μV
Ocular Vestibular Evoked Myogenic Potential (oVEMP): | Measured at baseline.
  Outcome measures: left-right asymmetry ratio in percent (%)
Computerized Dynamic Posturography (CDP) | Measured at baseline.
  Outcome measures: Sensory Organization Test (SOT):
  * Average equilibrium score (ES) for SOT1-6. Equilibrium scores is the average of three trials for each of the six conditions SOT1-6.
  * The SOT Composite score. It is a weighted average of the six conditions (SOT1-6) with greater weight given to the more difficult conditions.
  * The preference score. The preference score = (SOT3 + SOT6) / (SOT2 + SOT5)).
Computerized Dynamic Posturography (CDP) | Measured at baseline.
  Outcome measures: Motor Control Test (MCT):
  • Mean latency of the medium and the big movement respectively in anterior and posterior direction measured in milliseconds.
Computerized Dynamic Posturography (CDP) | Measured at baseline.
  Outcome measures: ADaptation Test (ADT):
  • Mean sway energy score of toes-up and toes-down respectively. The sway energy score quantifies the force magnitude required to overcome the postural instability.

SECONDARY OUTCOMES:
Vestibular dysfunction | Measures at baseline
  Prevalence of vestibular dysfunction
Dizziness Handicap Inventory for patient caregivers (DHI-PC): | Measured at baseline.
  Outcome measures: Mean total DHI-PC score. DHI-PC is a caregiver-reported 21-item questionnaire. For each question there are three possible answers: yes, sometimes or no. Each answer provides respectively 4, 2 and 0 points. The total DHI scores range from 0 to 84 with higher score being consistent with more limitation and more severe handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Therese Ovesen, Professor, Study Chair — University Clinic for Balance, Flavour and Sleep, Department of ENT, Gødstrup Hospital, DK
Locations (1):
- Gødstrup Regional Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No